CLINICAL TRIAL: NCT03104452
Title: Enhancing the Delivery of Tobacco Treatment During Pregnancy and Postpartum Though Systems-Change
Brief Title: Helping Moms Who Smoke
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: K01DA040745 (NIH)
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Smokers: Participants are pregnant women who smoked in the six months prior to their pregnancy.

SUMMARY:
The purpose of this study is to learn how women's smoking changes during their pregnancy and as a new mom, and to assess the help they receive from their health care providers.

DETAILED DESCRIPTION:
Approximately 90% of women who smoked before pregnancy will be smokers within one year of delivery . This occurs even though half who smoke quit during the course of pregnancy. This is an observational, cohort study of pregnant women who smoked in the six months before becoming pregnant. Women will be followed from the first trimester to one year after the birth of their babies. The results of this study will help us to describe women's' views on the quality of tobacco counseling they receive from their doctors; understand patterns of smoking and quitting throughout pregnancy and after childbirth; and provide information needed to develop an intervention to help women quit.

ELIGIBILITY:
Inclusion Criteria:

* Smoked within six months prior to becoming pregnant or current smoking
* Smoked at least 100 cigarettes
* Pregnant
* English speaking
* Access to a cell phone
* Willing to receive and send text messages.

Exclusion Criteria:

* Quit for longer than 6 months before becoming pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women will be included in this study.
Study Population: Participants will be recruited from obstetric and family practice clinics identified by the researchers.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Smoking status | 1 year post-partum
  The investigators will assess 7-day point prevalence smoking status over multiple time-points over the study period

CONTACTS AND LOCATIONS:
Overall Officials: Taneisha Scheuermann, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No